CLINICAL TRIAL: NCT04186299
Title: The Effect of Buccal Infiltration Administration of Clonidine on the Success Rate of Inferior Alveolar Nerve Block on Mandibular Molars With Symptomatic Irreversible Pulpitis: a Randomized Double-blind Clinical Trial
Brief Title: The Effect of Buccal Infiltration Administration of Clonidine on the Success Rate of Inferior Alveolar Nerve Block
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study activities never commenced.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-28605
Record Dates: First submitted 2019-11-21; First posted 2019-12-04 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Clonidine; Carticaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clonidine + articaine/epinephrine (Experimental): 1.7mL of 4% articaine/epinephrine(1:100,000) + clonidine (15ug/ml)
  Interventions: Drug: Clonidine; Drug: Articaine Hydrochloride + Epinephrine
- articaine/epinephrine (Active Comparator): 1.7mL of 4% articaine with 1:100,000 epinephrine
  Interventions: Drug: Articaine Hydrochloride + Epinephrine

INTERVENTIONS:
Drug: Clonidine — Each patient will receive a buccal infiltration of 1.7mL of 1:100,000 clonidine.
  Arms: Clonidine + articaine/epinephrine
Drug: Articaine Hydrochloride + Epinephrine — Each patient will receive a buccal infiltration of 1.7mL of 4% articaine with 1:100,000 epinephrine.

SUMMARY:
Articaine/epinephrine and lidocaine/epinephrine are the most common routine local anesthetic agents currently used in dentistry. However, their anesthetic efficacy and pain control in patients with symptomatic irreversible pulpitis via inferior alveolar nerve block is very low. The aim of this study is to investigate the efficacy of clonidine versus articaine/epinpephrine as a local anesthetic agent for a buccal infiltration after IANB administration with lidocaine for (1) successful IANB, (2) hemodynamic stability, and (3) reducing dental anxiety for endodontic treatment in mandibular molars diagnosed with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Articaine/epinephrine and lidocaine/epinephrine are the most common routine local anesthetic agents currently used in dentistry. However, their anesthetic efficacy and pain control in patients with symptomatic irreversible pulpitis via inferior alveolar nerve block is very low. The aim of this study is to investigate the efficacy of clonidine versus articaine/epinpephrine as a local anesthetic agent for a buccal infiltration after IANB administration with lidocaine for (1) successful IANB, (2) hemodynamic stability, and (3) reducing dental anxiety for endodontic treatment in mandibular molars diagnosed with symptomatic irreversible pulpitis. 100 patients with first or second mandibular molars diagnosed with symptomatic irreversible pulpitis will be enrolled. Patients will randomly receive either 1.7mL of clonidine (1:100,000) or 1.7mL of 4% articaine with epinephrine (1:100,000) using buccal infiltration technique after administration of 1.7mL of 2% lidocaine with epinephrine (1:100,000) using an IANB technique. 15 minutes after injection, lip numbness will be checked. Those who reported lip numbness will be checked for pulpal anesthesia. Those who achieve profound pulpal anesthesia will be included in the study. Patient's pain score will be recorded using a Heft-Parker visual analog scale before, during and after endodontic treatment. Success in IANB is defined as no or mild pain upon endodontic access cavity preparation and initial canal instrumentation. The hemodynamic parameters and pain management will be measured before and after root canal treatment with specific intervals. Patient's dental anxiety level will be measured by VAS-Anxiety preoperatively, before IANB administration, before endodontic treatment and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Must be in general good health as determined by the Investigator based on a review of the health history/update for participation in the trial (American Society of Anesthesiologists classification 1); and
* Have a diagnosis of symptomatic irreversible pulpitis and symptomatic apical periodontitis for their mandibular first or second molar.

Exclusion Criteria:

* Active signs of oral infections or inflammation;
* History of addiction or use of beta blockers;
* Use of medications that could affect anesthetic assessment (opioids at least one week before treatments);
* Allergies or contraindications to the use of clonidine, epinephrine or ibuprofen;
* Pregnant or nursing per subject report;
* No response to cold testing;
* Any diseases or condition that might interfere with the safe participation in the study; and
* Inability to undergo study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of success of IANB | The pain level is recorded as the extent of access is achieved within dentin and while entering the pulp chamber or during initial file placement. Data of each patient will be recorded through study completion, an average of 4 hours.
  The patients will be instructed to rate any pain felt during the procedure. If they feel pain, the treatment will be stopped immediately and they rate their pain using the Heft-Parker Visual Analogue Scale (VAS). The success of the IANB is defined as the ability to penetrate dentin, enter the pulp and advance instruments into the coronal part of the canal pulp without pain or with mild pain. The VAS consists of four categories of scales on a 170mm VAS line. No pain corresponds to 0mm. Mild pain is defined as greater than 0mm and less than or equal to 54mm. Moderate pain is defined as greater 54mm and less than or equal to 114mm. Severe pain is defined as greater than 114mm. At each step, when patients report moderate to severe pain, the IANB is considered to have failed.

SECONDARY OUTCOMES:
Evaluation of dental anxiety | The initial measurement is obtained before treatment, and 5 and 30 minutes after administration of anesthesia. Data of each patient are recorded by the end of the visit, which takes an average of 4 hours.
  Patients are instructed to rate their dental anxiety level on a VAS-Anxiety. The VAS consists of four categories of scales on a 10cm VAS line. No anxiety corresponds to 0cm. Mild anxiety is defined as greater than 0cm and less than 5.1cm. Moderate anxiety is defined as greater than or equal to 5.1cm and less than 7.0cm. Severe anxiety is defined as greater than or equal to 7.0cm.

CONTACTS AND LOCATIONS:
Overall Officials: Elham Shadmehr, DDS, MS, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No